CLINICAL TRIAL: NCT07335653
Title: A Randomized Controlled Trial Evaluating High-Purity Type I Collagen Wrap Around Extensor Tendon Repair Sites in Zones VI-VIII of the Hand to Prevent Adhesions and Improve Functional Outcomes
Brief Title: Evaluation of High-Purity Type I Collagen Biologic Wrap to Improve Function After Extensor Tendon Repair of the Hand
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Collaborators: Mysore Medical College and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIMS/IEC/270/2025
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Injury of Extensor Tendon of Hand; Tendon Adhesions
Keywords: Extensor tendon repair; Tendon adhesion; High Purity Type I Collagen; Biologic wrap; Hand injuries
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPTC Wrap + Standard Extensor Tendon Repair (Active Comparator): After completion of standard extensor tendon repair, a sterile high-purity Type I collagen sheet is hydrated, trimmed, and loosely wrapped circumferentially around the repaired tendon segment to act as a resorbable biologic barrier aimed at reducing peritendinous adhesions.
  Interventions: Device: High-Purity Type I Collagen (HPTC) Wrap; Procedure: Standard Extensor Tendon Repair
- Standard Extensor Tendon Repair Alone (Other): Primary extensor tendon repair using standard core and epitendinous sutures without use of any biologic wrap or anti-adhesion adjunct.
  Interventions: Procedure: Standard Extensor Tendon Repair

INTERVENTIONS:
Device: High-Purity Type I Collagen (HPTC) Wrap — After completion of standard extensor tendon repair, a sterile high-purity Type I collagen sheet is hydrated, trimmed, and loosely wrapped circumferentially around the repaired tendon segment to act as a resorbable biologic barrier aimed at reducing peritendinous adhesions.
  Arms: HPTC Wrap + Standard Extensor Tendon Repair
Procedure: Standard Extensor Tendon Repair — Primary extensor tendon repair using standard core and epitendinous sutures without use of any biologic wrap or anti-adhesion adjunct.

SUMMARY:
Tendon injuries of the hand, particularly extensor tendons, are prone to postoperative adhesions, extensor lag, and stiffness, leading to functional impairment. This multicentric randomized controlled trial evaluates whether wrapping repaired extensor tendons with a high-purity Type I collagen (HPTC) biologic membrane can reduce adhesion formation and improve functional outcomes compared with standard repair alone.

DETAILED DESCRIPTION:
Extensor tendon injuries of the hand are common due to the superficial location of the tendons and the thin soft tissue envelope over the dorsum of the hand and wrist. These injuries, particularly in zones VI-VIII, are frequently associated with postoperative adhesions and extensor lag, leading to functional impairment and delayed return to work. Postsurgical adhesions may occur in up to 30-40% of tendon injuries and remain a major clinical challenge despite advances in suture techniques and rehabilitation protocols.

Several strategies have been investigated to minimize tendon adhesions, including optimized suture techniques, early mobilization, anti-adhesive agents, and biologic barrier membranes. Recent clinical work has shown that wrapping repaired extensor tendons with an amniotic membrane in zone VI can improve range of motion (ROM), Quick DASH scores, and recovery time, suggesting a true reduction in peritendinous fibrosis. Experimental models have also demonstrated that collagen-glycosaminoglycan (GAG) wraps can reduce early postoperative tendon adhesions while preserving tendon healing strength.

HPTC is a bioengineered, acellular dermal replacement product composed of >97% pure Type I collagen, free of elastin, lipids, and immunogenic proteins. It is manufactured to preserve the native triple helical structure and bioactivity of collagen, providing a cell-conducive scaffold that promotes neovascularization, granulation tissue formation, and tissue remodelling. HPTC is flexible, translucent, moderately tacky, and can be cut, sutured or stapled, making it feasible to be fashioned as a wrap or sleeve around tendons.

Multiple randomized controlled trials and clinical series by Narayan et al. have demonstrated the safety and efficacy of high-purity Type I collagen-based skin substitute HPTC in chronic and acute wounds.

These studies collectively show that high-purity Type I collagen membranes are safe, well tolerated, promote faster wound healing, and have favourable scarring and pain profiles in a variety of clinical settings.

Rationale for the Current Study - Given the strong biological plausibility of Type I collagen scaffolds as biocompatible, resorbable barriers that can modulate the healing milieu; the safety and clinical efficacy of HPTC in multiple wound types; and the demonstrated benefit of biologic wraps (e.g., amniotic membrane) around extensor tendon repairs in reducing adhesions, it is logical to evaluate whether a HPTC wrap around the repaired extensor tendon in zones VI-VIII can reduce adhesion-related stiffness and improve functional outcomes compared with standard repair alone.

This trial will be, to our knowledge, the first prospective randomized clinical trial to assess HPTC as a tendon wrap in extensor tendon repairs of the hand.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Acute open laceration of extensor tendons in zone VI, VII, or VIII of the hand / wrist (according to Verdan's classification), involving digits 2-5 and/or wrist extensors.
3. Complete tendon laceration (≥50% tendon cross-sectional area), requiring primary repair.
4. Time from injury to surgical repair ≤72 hours.
5. Single upper limb involved.
6. Ability and willingness to comply with postoperative rehabilitation protocol and follow-up visits.
7. Provision of written informed consent.

Exclusion Criteria:

1. Crush, avulsion, or segmental tendon loss requiring graft or tendon transfer.
2. Associated open fractures requiring dorsal plating across the repair site, or extensive bone loss affecting joint stability.
3. Previous surgery or significant scarring over the injured extensor tendon region.
4. Associated major nerve injury requiring graft or complex reconstruction (digital nerve repair without grafting may be allowed if balanced between groups).
5. Uncontrolled systemic illness (e.g., HbA1c > 8.5% for diabetes, severe peripheral vascular disease, chronic steroid use, severe malnutrition).
6. Active infection at the injury site.
7. Known allergy or hypersensitivity to bovine/ovine collagen or any component of HPTC.
8. Pregnancy or lactation.
9. Inability to provide informed consent or comply with follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Total Active Motion (TAM) of Involved Finger(s) | 8 weeks postoperatively
  Total Active Motion (TAM) is calculated as the sum of active flexion at the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints minus the extension deficits. TAM is expressed in degrees and as a percentage of the contralateral uninvolved digit or standard normative values. Higher values indicate better functional outcome.

SECONDARY OUTCOMES:
QuickDASH Score | 6 weeks and 8 weeks postoperatively
  Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire assessing upper limb disability and symptoms. Lower scores indicate better function.
Extensor Lag | 8 weeks postoperatively
  Measured as the deficit in active extension at MCP, PIP, and DIP joints compared with neutral position and the contralateral side.
Adhesion-Related Events | Up to 8 weeks postoperatively
  Clinically significant adhesions defined as failure to achieve Total Active Motion ≥60% by 8 weeks despite compliant therapy and/or requirement for surgical tenolysis.
Grip Strength | 8 weeks postoperatively
  Measured using a calibrated Jamar dynamometer and expressed as absolute values and percentage of the contralateral side.
Complication Rates | From surgery to 8 weeks postoperatively
  Incidence of wound infection, wound dehiscence, tendon re-rupture, hypersensitivity reactions, foreign body response, and complex regional pain syndrome.
Time to Return to Work or Activities of Daily Living | Up to 8 weeks postoperatively
  Number of days from surgery to return to pre-injury occupational or activities of daily living status.
Patient Satisfaction | 8 weeks postoperatively
  Patient-reported satisfaction with hand function and appearance measured using Likert scale. Scale range: 1 to 5 (1 = very dissatisfied, 5 = very satisfied). Interpretation: Higher scores indicate greater patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (2):
- India (2):
  - Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in the primary and secondary outcome analyses will be shared. This includes demographic variables, injury characteristics, intervention allocation, Total Active Motion (TAM) measurements, QuickDASH scores, extensor lag measurements, grip strength values, complication data, and time-to-return-to-work variables. Data dictionaries and metadata necessary to interpret the shared datasets will also be provided.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available beginning 6 months after publication of the primary study results and will remain available for a period of 5 years following publication.
Access Criteria: IPD will be shared with qualified researchers who submit a methodologically sound research proposal and agree to the terms of data use.
  IPD may be used for meta-analyses, secondary analyses, methodological research, or validation studies related to tendon repair outcomes and adhesion prevention strategies.
  Data will be shared upon reasonable request through secure institutional data-sharing platforms or encrypted electronic transfer after execution of a data use agreement (DUA). All shared data will be fully de-identified to protect participant confidentiality, in accordance with applicable ethical and regulatory guidelines.

REFERENCES:
- [Background] 15. Wong JKF, Metcalfe AD, Wong R, Bush J, Platt C, McGrouther DA. Reduction of tendon adhesion formation with a collagen-GAG scaffold: an experimental study. J Hand Surg Eur Vol. 2006;31(2):143-150.
- [Background] Moran SL, Ryan CK, Orlando GS, Ehara K, Hentz VR. Effects of anti-adhesion barriers on the healing of repaired extensor digitorum communis tendons in a rabbit model. J Hand Surg Am. 2000;25(3):546-553.
- [Background] Narayan N, Raghupathi D, Ramamurthy V, Chethan S, Gowda S. A Comparative Analysis in the Treatment of Full-Thickness Wounds: Negative-Pressure Wound Therapy (NPWT) Combined With High-Purity Type I Collagen-Based Skin Substitute Versus NPWT Alone. Cureus. 2025 Nov 16;17(11):e96977. doi: 10.7759/cureus.96977. eCollection 2025 Nov. PMID 41250786
- [Background] Narayan N, Shivaiah R, Kumar V, Kumar KM, Chethan S, Gowda S. Comparative Efficacy of High Purity Type I Collagen-Based Skin Substitute and Dehydrated Human Amnion/Chorion Membrane in Diabetic Foot Ulcers: A Multicentre Randomized Controlled Trial. Cureus. 2025 Oct 19;17(10):e94952. doi: 10.7759/cureus.94952. eCollection 2025 Oct. PMID 41122365
- [Background] Narayan N, Ramegowda YH, Raghupathi DS, Chethan S, Gowda S. Biological Skin Substitutes in Pressure Ulcers: High-Purity Type I Collagen-Based Versus Amnion/Chorion Membrane. Cureus. 2025 Aug 25;17(8):e90956. doi: 10.7759/cureus.90956. eCollection 2025 Aug. PMID 40862036
- [Background] Narayan N, Shivannaiah C, Gowda S. Evaluating the Efficacy of High-Purity Type I Collagen-Based Skin Substitute Versus Dehydrated Human Amnion/Chorion Membrane in the Treatment of Venous Leg Ulcers: A Randomized Controlled Clinical Trial. Cureus. 2025 Jul 30;17(7):e89031. doi: 10.7759/cureus.89031. eCollection 2025 Jul. PMID 40747200
- [Background] Wong JK, Lui YH, Kapacee Z, Kadler KE, Ferguson MW, McGrouther DA. The cellular biology of flexor tendon adhesion formation: an old problem in a new paradigm. Am J Pathol. 2009 Nov;175(5):1938-51. doi: 10.2353/ajpath.2009.090380. Epub 2009 Oct 15. PMID 19834058
- [Background] Al-Qattan MM. Controlled active motion following extensor tendon repair in zones V-VIII. J Hand Surg Br. 2005;30(2):166-169.
- [Background] VERDAN CE. Primary repair of flexor tendons. J Bone Joint Surg Am. 1960 Jun;42-A:647-57. No abstract available. PMID 13855215
- [Background] Newport ML, Blair WF, Steyers CM Jr. Long-term results of extensor tendon repair. J Hand Surg Am. 1990 Nov;15(6):961-6. doi: 10.1016/0363-5023(90)90024-l. PMID 2269792